CLINICAL TRIAL: NCT01258231
Title: Identification of Genomic Predictors of Adverse Events After Cardiac Surgery
Acronym: CABGGenomics
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Texas Heart Institute (Other); University of Texas Southwestern Medical Center (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jochen Daniel Muehlschlegel, MD, Professor, Johns Hopkins University
Other Study IDs: 2000P001639; 5R01HL098601 (NIH); NCT00281164 (obsolete NCT alias)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Genetic Predisposition to Disease; Atrial Fibrillation; Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Genetic Predisposition to Disease; Atrial Fibrillation; Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, buffy coat, plasma, serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery: Adult patients undergoing cardiac surgery

SUMMARY:
This study aims to identify genetic causes of adverse events after cardiac surgery, such as atrial fibrillation, myocardial infarction, renal dysfunction and heart failure.

Patients undergoing heart surgery at Brigham and Women's Hospital and Texas Heart Institute are eligible to participate.

DETAILED DESCRIPTION:
This study aims to identify genetic causes of adverse events after cardiac surgery, such as atrial fibrillation, myocardial infarction, renal dysfunction and heart failure. In addition, we also examine blood and urine biomarkers (proteins).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing heart surgery
* Willing to provide consent

Exclusion Criteria:

* Enrolled in a concurrent drug or device trial that precludes concurrent enrollment

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2000-08 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Mortality (i.e. number of participants who are deceased during postoperative day 0 up to year 5) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include serum creatinine.

OTHER OUTCOMES:
Acute Kidney Injury using KDIGO criteria: albumin/creatinine ratio (>/= 300 mg/g) and eGRF (< 60 mL/min/1.73^2) | Day of procedure to post procedure day 7
  Data will be collected from electronic medical records; data points to be collected for this measurement include serum creatinine.
Presence of Arrhythmia (i.e. number of patients who develop an arrhythmia after their cardiac surgery) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post-procedural EKG reports and progress notes.
Myocardial Infarction (i.e. number of participants who develop a MI during postoperative day 0 to year 5) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post-procedural EKG reports, cardiac enzyme values, progress notes, and cardiac catheterization reports.
Heart failure per NYHA class II, III, IV | Day of procedure to year 5
  This will be measured in accordance to New York Heart Association Guidelines.
Quality of Life Survey - The Kansas City Cardiomyopathy Questionnaire (KCCQShortForm) | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  A questionnaire to assess for heart failure
Quality of Life Survey - The Seattle Angina Questionnaire (SAQShortForm) | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  A questionnaire to assess for angina
Quality of Life Survey - 12-item short form health survey (SF12) | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  A questionnaire to assess for overall health

CONTACTS AND LOCATIONS:
Overall Officials: Jochen D Muehlschlegel, MD MMSc, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UT Southwestern Medical Center, Dallas, Texas
  - Department Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas

REFERENCES:
- [Background] Sigurdsson MI, Muehlschlegel JD, Fox AA, Heydarpour M, Lichtner P, Meitinger T, Collard CD, Shernan SK, Body SC. Genetic Variants Associated With Atrial Fibrillation and PR Interval Following Cardiac Surgery. J Cardiothorac Vasc Anesth. 2015;29(3):605-10. doi: 10.1053/j.jvca.2014.10.028. Epub 2014 Nov 4. PMID 26009287
- [Background] Barnet CS, Liu X, Body SC, Collard CD, Shernan SK, Muehlschlegel JD, Jarolim P, Fox AA. Plasma corin decreases after coronary artery bypass graft surgery and is associated with postoperative heart failure: a pilot study. J Cardiothorac Vasc Anesth. 2015 Apr;29(2):374-81. doi: 10.1053/j.jvca.2014.11.001. Epub 2014 Nov 11. PMID 25649697
- [Background] Fox AA, Pretorius M, Liu KY, Collard CD, Perry TE, Shernan SK, De Jager PL, Hafler DA, Herman DS, DePalma SR, Roden DM, Muehlschlegel JD, Donahue BS, Darbar D, Seidman JG, Body SC, Seidman CE. Genome-wide assessment for genetic variants associated with ventricular dysfunction after primary coronary artery bypass graft surgery. PLoS One. 2011;6(9):e24593. doi: 10.1371/journal.pone.0024593. Epub 2011 Sep 30. PMID 21980348
- [Background] Fox AA, Marcantonio ER, Collard CD, Thoma M, Perry TE, Shernan SK, Muehlschlegel JD, Body SC. Increased peak postoperative B-type natriuretic peptide predicts decreased longer-term physical function after primary coronary artery bypass graft surgery. Anesthesiology. 2011 Apr;114(4):807-16. doi: 10.1097/ALN.0b013e31820ef9c1. PMID 21427536
- [Background] Muehlschlegel JD, Liu KY, Perry TE, Fox AA, Collard CD, Shernan SK, Body SC; CABG Genomics Investigators. Chromosome 9p21 variant predicts mortality after coronary artery bypass graft surgery. Circulation. 2010 Sep 14;122(11 Suppl):S60-5. doi: 10.1161/CIRCULATIONAHA.109.924233. PMID 20837927
- [Background] Muehlschlegel JD, Perry TE, Liu KY, Fox AA, Collard CD, Shernan SK, Body SC. Heart-type fatty acid binding protein is an independent predictor of death and ventricular dysfunction after coronary artery bypass graft surgery. Anesth Analg. 2010 Nov;111(5):1101-9. doi: 10.1213/ANE.0b013e3181dd9516. Epub 2010 May 10. PMID 20457766
- [Background] Perry TE, Muehlschlegel JD, Liu KY, Fox AA, Collard CD, Shernan SK, Body SC; CABG Genomics Investigators. Plasma neutrophil gelatinase-associated lipocalin and acute postoperative kidney injury in adult cardiac surgical patients. Anesth Analg. 2010 Jun 1;110(6):1541-7. doi: 10.1213/ANE.0b013e3181da938e. Epub 2010 Apr 30. PMID 20435938
- [Background] Perry TE, Muehlschlegel JD, Liu KY, Fox AA, Collard CD, Body SC, Shernan SK; CABG Genomics Investigators. Preoperative C-reactive protein predicts long-term mortality and hospital length of stay after primary, nonemergent coronary artery bypass grafting. Anesthesiology. 2010 Mar;112(3):607-13. doi: 10.1097/ALN.0b013e3181cea3b5. PMID 20179497
- [Background] Garvin S, Muehlschlegel JD, Perry TE, Chen J, Liu KY, Fox AA, Collard CD, Aranki SF, Shernan SK, Body SC. Postoperative activity, but not preoperative activity, of antithrombin is associated with major adverse cardiac events after coronary artery bypass graft surgery. Anesth Analg. 2010 Oct;111(4):862-9. doi: 10.1213/ANE.0b013e3181b7908c. Epub 2009 Oct 9. PMID 19820236
- [Background] Perry TE, Muehlschlegel JD, Liu KY, Fox AA, Collard CD, Body SC, Shernan SK; CABG Genomics Investigators. C-Reactive protein gene variants are associated with postoperative C-reactive protein levels after coronary artery bypass surgery. BMC Med Genet. 2009 May 8;10:38. doi: 10.1186/1471-2350-10-38. PMID 19426506
- [Background] Muehlschlegel JD, Perry TE, Liu KY, Nascimben L, Fox AA, Collard CD, Avery EG, Aranki SF, D'Ambra MN, Shernan SK, Body SC; CABG Genomics Investigators. Troponin is superior to electrocardiogram and creatinine kinase MB for predicting clinically significant myocardial injury after coronary artery bypass grafting. Eur Heart J. 2009 Jul;30(13):1574-83. doi: 10.1093/eurheartj/ehp134. Epub 2009 Apr 30. PMID 19406870
- [Derived] Body SC, Collard CD, Shernan SK, Fox AA, Liu KY, Ritchie MD, Perry TE, Muehlschlegel JD, Aranki S, Donahue BS, Pretorius M, Estrada JC, Ellinor PT, Newton-Cheh C, Seidman CE, Seidman JG, Herman DS, Lichtner P, Meitinger T, Pfeufer A, Kaab S, Brown NJ, Roden DM, Darbar D. Variation in the 4q25 chromosomal locus predicts atrial fibrillation after coronary artery bypass graft surgery. Circ Cardiovasc Genet. 2009 Oct;2(5):499-506. doi: 10.1161/CIRCGENETICS.109.849075. Epub 2009 Aug 2. PMID 20031626